CLINICAL TRIAL: NCT05579054
Title: Translation, Validity, and Reliability of the Foot Posture Index (FPI-6) - Turkish Version
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Gullu Aydın Yagcıoglu, Research Asisstant, Suleyman Demirel University
Other Study IDs: FPI-6
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Foot Deformities; Pes Planus; Hallux Valgus; Metatarsalgia; Feet Pes Planus (Flatfoot)
MeSH Terms: conditions — Foot Deformities; Flatfoot; Hallux Valgus; Metatarsalgia; Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Foot Posture Index (FPI-6) — FPI-6 is a valid and reliable assessment tool for pediatrics in which 6 items are scored separately for the right and left feet while the patient was in an upright position in a relaxed posture with their body-weight evenly distributed on the both feet. Each item is scored as -2, -1, 0, 1, 2 and the assessment categorized as follows: 0 to +5 normal; +6 to +9 pronated; 10+ higly pronated; -1 to -4 supianted; and -5 to -12 higly supinated.

SUMMARY:
Individuals with foot-ankle problems (plantar fasciitis, metarsalgia, pes planus, pes planovalgus/varus) will be included in the study. Permission was obtained from the research group that developed the scale to use the Original Foot Posture Index-6 (FPI-6). Cross-cultural adaptation of the FPI-6 will be made in line with the guidelines published by Ruberto and Beaton. First of all, the FPI-6 will be translated into Turkish by two translators whose native language is Turkish and who can speak English at an advanced level. Translations will be compared and discussed, and a Turkish version will be obtained with the equivalents that best represent each item in the texts. Secondly, this retranslated text will be independently translated back into English by two native English translators. In the third stage, two texts written in English will be synthesized by the authors, thus reaching a consensus on a single translation. Finally, the inconsistent parts of the text will be checked by a multidisciplinary team consisting of two native English-speaking translators, members of the English language and literature department, authors who developed the scale, and physiotherapists. Two independent physiotherapists will evaluate the participants' foot posture indexes by FPI-6 for inter-rater reliability. In addition, patients' quality of life, foot functions, hindfoot profiles will be evaluated. For the calculation of validity between measurements, rater-1 will apply the FPI-6 again to the same participants after 15 days for intra-rater reliability. Patients' functional independence, activities of daily living, and quality of life will also be evaluated for criterion validity. American Orthopedic Foot and Ankle Society-AOFAS, SF-36 and Foot Function Index questionnaires will be applied for the validity of FPI-6.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18-65,
* having foot-ankle problems (plantar fasciitis, metatarsalgia, pes planus, pes planovalgus/varus, hallux valgus, pes cavus, pain)

Exclusion Criteria:

* Having undergone any lower extremity surgery in the last two years,
* patients with congenital foot deformity and neurological problems,
* Individuals with lower or upper extremity pathology or a cognitive problem that may prevent or limit the application of the test protocol

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study group will consist of individuals between the ages of 18-65 with foot problems.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Foot Posture Index (FPI-6) | 10 minutes
  PI-6 is a valid and reliable assessment tool for pediatrics in which 6 items are scored separately for the right and left feet while the patient was in an upright position in a relaxed posture with their body-weight evenly distributed on the both feet. Each item is scored as -2, -1, 0, 1, 2 and the assessment categorized as follows: 0 to +5 normal; +6 to +9 pronated; 10+ higly pronated; -1 to -4 supianted; and -5 to -12 higly supinated.

SECONDARY OUTCOMES:
Foot Function Index | 10 minutes
  Foot Function Index consists of 23 items with 3 subgroups as pain, disability and activity limitation. While the nine-item pain subscale measures the level of foot pain in various situations, the 9-item disability subscale determines the degree of difficulty in performing various functional activities depending on foot problems.
American Orthopedic Foot and Ankle Society-AOFAS | 10 minutes
  American Orthopedic Foot and Ankle Society-AOFAS; This method, which evaluates the foot alignment and functional status of the participants, is the valid and reliable scoring system of the Turkish version developed by the American Foot and Ankle Orthopedic Society. The pain subscale is evaluated over a total of 40 points, the function subscale is evaluated over a total of 50 points, and the foot alignment subscale is evaluated over a total of 10 points. Higher scores indicate a better situation.
SF-36 | 15 minutes
  The SF-36 QoL test includes a total of 36 self-assessment questions that are classified into eight domains: physical functioning with ten questions, role-physical with four, bodily pain with two, general health with five, social functioning with two, role-emotional with three, mental health with five and vitality with four. The reference period for all of the questions was the last four weeks prior to the interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Güllü Aydın Yağcıoğlu, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided